CLINICAL TRIAL: NCT05772975
Title: Evaluation of Soft and Hard Tissue Healing After Impacted Mandibular Third Molar Surgery With the Use of E-PRF and H-PRF - a Randomized Controlled Clinical Study
Brief Title: The Clinical Impact of E-PRF and H-PRF on Healing After Mandibular Third Molar Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amila Haskic (Other)
Responsible Party: Sponsor-Investigator, Amila Haskic, Principal Investigator, University of Sarajevo
Organization: University of Sarajevo (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 02-3-4-59-1-3/2021
Record Dates: First submitted 2023-02-15; First posted 2023-03-17 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Platelet-Rich Fibrin
Keywords: Molar, Third; PRF; Platelet-Rich Fibrin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- E-PRF (Experimental): After the impacted mandibular third molar has been surgically removed E-PRF is placed in the dentoalveolar defect and the wound is primarily closed.
  Interventions: Biological: E-PRF
- H-PRF (Experimental): After the impacted mandibular third molar has been surgically removed H-PRF is placed in the dentoalveolar defect PRF made with horizontal centrifuge and the wound is primarily closed.
  Interventions: Biological: H-PRF (Horizontal-platelet rich fibrin)
- CONTROL (No Intervention): After the impacted mandibular third molar has been surgically removed, the wound is primarily closed.

INTERVENTIONS:
Biological: H-PRF (Horizontal-platelet rich fibrin) — Platelet-rich fibrin is an autologous biomaterial originating from human blood following centrifugation without additives that contains supraphysiological doses of growth factors. it serves as a biological healing matrix by supporting cell migration and cytokine release. H-PRF is obtained by horizontal centrifugation using (Bio-PRF) centrifuge on 700 g force for 8 minutes. This way the cells separate much more efficiently throughout the entire membrane/clot.
  Arms: H-PRF
Biological: E-PRF — Platelet-rich fibrin is an autologous biomaterial originating from human blood following centrifugation without additives that contains supraphysiological doses of growth factors. In order to extend its resorption period heating method is used. After centrifugation of blood using (Bio-PRF) centrifuge on 700 g force for 8 minutes top layer is heated for 10 minutes at 75°C in BIO-Heat device. When cooled it is mixed with cell rich buffy coat. This way PRF with extended life is obtained.
  Arms: E-PRF

SUMMARY:
This clinical trial aims to compare the effect of platelet concentrates E-PRF and H-PRF on soft and hard tissue healing in healthy individuals after lower third molar surgery. The main questions it aims to answer are:

Do E-PRF and H-PRF reduce complications after third molar surgery? Do E-PRF and H-PRF improve soft tissue healing after third molar surgery? Do E-PRF and H-PRF improve hard tissue healing after third molar surgery? Participants will be divided into 2 study groups and one control group. Third molar surgery will be performed according to standard protocol. In study groups, dentoalveolar defects will be filled with E-PRF and H-PRF which are products of centrifugation of the patient's blood without additives. Soft tissue and hard tissue healing will be compared between the groups.

DETAILED DESCRIPTION:
A Randomized, Three Parallel Arms Clinical Trial. The primary objective is to assess the clinical impact of E-PRF vs H-PRF vs Control on the soft tissue healing and post-op discomfort and complications after mandibular third molar surgery between the three groups during the healing period of 7 days.

The secondary objective is to compare bony healing between the three groups over three months using an Orthopantomograph (OPG) X-ray.

All subjects from the University of Sarajevo Faculty of Dentistry with Dental Clinical Center. Subjects that are coming for the removal of impacted mandibular third molars and match the inclusion criteria will be told about the research and offered the opportunity to participate.

ELIGIBILITY:
Inclusion Criteria:

* Orthodontic indication for impacted mandibular third molar surgery
* Physical status I according to the guidelines of the American Society of Anesthesiologists (ASA)

Exclusion Criteria:

* Presence of systemic disease
* Presence of a condition that affects fibrin clot formation
* History of radiation therapy or chemotherapy
* Allergy to penicillin
* Oral contraceptive usage
* Smoking habit
* Status of pregnancy or lactation
* Presence of any acute local infection
* Missing the adjacent second molar or indicated for extraction

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 61 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
The impact of E-PRF vs H-PRF vs Control on soft tissue healing | 3 days
  Soft tissue healing evaluation will be done by modified Landry, Turnbull and Howley healing index. For each post-extraction site, the following parameters will be evaluated by dichotomic scale (0/1): tissue color, response to palpation, presence of granulation tissue, epithelialization of incision margins and suppuration.
The impact of E-PRF vs H-PRF vs Control on soft tissue healing | 7 days
  Soft tissue healing evaluation will be done by modified Landry, Turnbull and Howley healing index. For each post-extraction site, the following parameters will be evaluated by dichotomic scale (0/1): tissue color, response to palpation, presence of granulation tissue, epithelialization of incision margins and suppuration.
The impact of E-PRF vs H-PRF vs Control on bone regeneration | 1 month
  Bone healing will be evaluated by comparing digital OPGs i.e. radiographic bone densitiy profiles in extraction sockets will be compared.
The impact of E-PRF vs H-PRF vs Control on bone regeneration | 3 months
  Bone healing will be evaluated by comparing digital OPGs i.e. radiographic bone densitiy profiles in extraction sockets will be compared.

SECONDARY OUTCOMES:
The impact of E-PRF vs H-PRF vs Control on periodontal pocket depth | 1 month
  Pocket depth will be measured using a periodontal probe taken from the margin of the gingiva to the base of the pocket along the distal surface of the mandibular second molar at three points: distobuccal, mid-distal, distolingual- by a single evaluator. Periodontal pocket depth will be measured preoperatively, one month and three months postoperatively
The impact of E-PRF vs H-PRF vs Control on periodontal pocket depth | 3 months
  Pocket depth will be measured using a periodontal probe taken from the margin of the gingiva to the base of the pocket along the distal surface of the mandibular second molar at three points: distobuccal, mid-distal, distolingual.
The impact of E-PRF vs H-PRF vs Control on postoperative trismus | 3 days
  The primary outcome is to asses the percentage of trismus after mandibular third molar surgery in study groups vs control. Trismus will be measured as the distance between the upper right and lower right central incisors during maximum mouth opening using digital caliper.
The impact of E-PRF vs H-PRF vs Control on postoperative trismus | 7 days
  The primary outcome is to asses the percentage of trismus after mandibular third molar surgery in study groups vs control. Trismus will be measured as the distance between the upper right and lower right central incisors during maximum mouth opening using digital caliper.
The impact of E-PRF vs H-PRF vs Control on postoperative swelling | 3 days
  The primary outcome is to asses the percentage of swelling after mandibular third molar surgery in study groups vs control. Facial swelling will be evaluated by measuring 3 facial distances: from the tragus to pogonion (TPO), tragus to labial commissure (TCO), and angulus mandibulae to lateral canthus (ACA).
The impact of E-PRF vs H-PRF vs Control on postoperative swelling | 7 days
  The primary outcome is to asses the percentage of swelling after mandibular third molar surgery in study groups vs control. Facial swelling will be evaluated by measuring 3 facial distances: from the tragus to pogonion (TPO), tragus to labial commissure (TCO), and angulus mandibulae to lateral canthus (ACA).
The impact of E-PRF vs H-PRF vs Control on postoperative pain | 7 days
  The primary outcome is to asses the level of pain after mandibular third molar surgery in study groups vs control. A visual analog scale (VAS) will be used to evaluate postoperative pain. A 10-point VAS with a score of 0 equals "no pain" and 10 equals "very severe pain" will be used to asses subjective pain. Patients will be asked to record number of analgesic taken during the monitoring period of 7days.

CONTACTS AND LOCATIONS:
Overall Officials: Amila Haskic, Principal Investigator — University of Sarajevo
Locations (1):
- Faculty of Dentistry with Dental Clinical Center, Sarajevo, Federation of Bosnia and Herzegovina, Bosnia and Herzegovina

IPD SHARING:
Plan to Share IPD: No